CLINICAL TRIAL: NCT03685760
Title: Reiki Intervention for Seriously Ill Elders Intensive Care Unit (RISE-ICU)
Acronym: RISE-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017H0402; GRT00051029 (Other Grant/Funding Number: American Association of Critical Care Nurses)
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mechanical Ventilation Complication; Complementary Health Approach
Keywords: Mechanically Ventilated Older Adults; Reiki; Pain; Agitation; Delirium
MeSH Terms: conditions — Pain; Psychomotor Agitation; Delirium | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Three Group Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor are masked as well as all investigators except one co-investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): Reiki will be administered for 5 consecutive days even if the subject is transferred to the floor from the ICU. Thirty minutes before and after the daily Reiki, session, the bedside nurse will obtain a set of baseline vital signs (heart rate, respiratory rate, blood pressure; non-invasively) for safety monitoring data.
  Interventions: Other: Reiki therapy
- Sham Reiki (Sham Comparator): Sham Reiki will be administered for 5 consecutive days even if the subject is transferred to the floor from the ICU. Thirty minutes before and after the daily sham Reiki, session, the bedside nurse will obtain a set of baseline vital signs (heart rate, respiratory rate, blood pressure; non-invasively) for safety monitoring data.
  Interventions: Other: Sham Reiki
- Usual Care (No Intervention): Twice per day, 30 minutes apart, the bedside nurse will obtain a set of baseline vital signs (heart rate, respiratory rate, blood pressure; non-invasively) for safety monitoring data. Usual care will also involve a 5-day period.

INTERVENTIONS:
Other: Reiki therapy — Reiki, a complementary health approach where trained practitioners place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. Reiki therapists will administer the Reiki intervention (i.e., a 30-minute treatment in which the subject is lightly touched for 3 minutes at each of 10 standardized Reiki hand positions).
  Arms: Reiki
Other: Sham Reiki — Sham (pretend) Reiki therapists will administer the sham Reiki intervention (i.e., a 30-minute treatment in which the subject is lightly touched for 3 minutes at each of 10 standardized Reiki hand positions). Sham providers do not have Reiki training.
  Arms: Sham Reiki

SUMMARY:
The overall objective of this proposal is to demonstrate the feasibility of conducting a future large-scale, randomized controlled trial (RCT) to test whether Reiki is superior to sham Reiki and usual care when delivered to critically ill older adults who require mechanical ventilation (MV). Our three-arm, pilot RCT will include 45 subjects and their LARs (45) recruited from the Ohio State University Wexner Medical Center (OSU-WMC) intensive care units (ICUs) who are randomly allocated 1:1:1 to: 1) Reiki, 2) sham Reiki, or 3) usual care for 5 days or until the subject is discharged from the hospital or expires. The Investigators will perform interviews with the subjects' LARs upon study enrollment to determine the subjects preadmission physical, functional, and cognitive health status. Each subject will be assessed for pain, anxiety, and agitation and have their vital signs taken daily for 5 days using valid and reliable tools. Medical records will be used to record demographic and clinical characteristics. The Investigators will survey each subject and their LAR regarding their experiences with the Reiki, sham Reiki or usual care sessions. Reiki and sham Reiki will be administered for 5 consecutive days even if the subject is transferred to the floor from the ICU. Usual care will also involve a 5-day period. Study Arms. Reiki. Three professional Reiki therapists trained at Level 2 (intermediate) and with a minimum of 2 years of Reiki practice will administer the Reiki intervention. Sham Reiki. Three actors will administer sham Reiki. Usual Care. Subjects assigned to usual care will not receive Reiki or sham Reiki. The usual care group will undergo the same in-person symptom assessments and electronic health record (EHR) reviews as the Reiki and sham Reiki groups. Reiki therapy is not part of usual care in the participating ICUs. The knowledge gained from this study will contribute to a better understanding of how/if a nonpharmacologic intervention can reduce the symptoms experienced by critically ill older adults.

DETAILED DESCRIPTION:
The overall objective of this proposal is to demonstrate the feasibility of conducting a future large-scale, randomized controlled trial (RCT) to test whether Reiki is superior to sham Reiki and usual care when delivered to critically ill older adults who require mechanical ventilation (MV). Our three-arm, pilot RCT will include 45 subjects and their LARs (45) recruited from the Ohio State University Wexner Medical Center (OSU-WMC) intensive care units (ICUs) who are randomly allocated 1:1:1 to: 1) Reiki, 2) sham Reiki, or 3) usual care for 5 days or until the subject is discharged from the hospital or expires. The Investigators will perform interviews with the subjects' LARs upon study enrollment to determine the subjects preadmission physical, functional, and cognitive health status. Each subject will be assessed for pain, anxiety, and agitation and have their vital signs taken daily for 5 days using valid and reliable tools. Medical records will be used to record demographic and clinical characteristics. The Investigators will survey each subject and their LAR regarding their experiences with the Reiki, sham Reiki or usual care sessions. Reiki and sham Reiki will be administered for 5 consecutive days even if the subject is transferred to the floor from the ICU. Usual care will also involve a 5-day period. Study Arms. Reiki. Three professional Reiki therapists trained at Level 2 (intermediate) and with a minimum of 2 years of Reiki practice will administer the Reiki intervention. The Reiki intervention involves a 30-minute treatment in which the participant is lightly touched for 3 minutes at each of 10 standardized Reiki hand positions (eyes, temples, crown, back of head, thymus/lungs, abdomen, scapula, mid back, lower back, feet). Sham Reiki. Three actors matched for age and sex with the Reiki therapists will administer sham Reiki. Sham interventionists may not be providers of any touch therapy or bodywork modalities (e.g. Reiki, Therapeutic Touch, Healing Touch, general massage) nor may they be providers of any type of complementary therapies (e.g. aromatherapy, guided imagery, hypnosis). The sham Reiki session consists of 30-minutes of direct contact using the same 10 standardized hand positions as the Reiki intervention. To minimize unconscious healing intentions, sham interventionists will occupy their minds with thoughts unrelated to the participant (e.g., counting backwards from 100 to 1). Usual Care. Subjects assigned to usual care will not receive Reiki or sham Reiki. The usual care group will undergo the same in-person symptom assessments and electronic health record (EHR) reviews as the Reiki and sham Reiki groups. Reiki therapy is not part of usual care in the participating ICUs. The knowledge gained from this study will contribute to a better understanding of how/if a nonpharmacologic intervention can reduce the symptoms experienced by critically ill older adults.

ELIGIBILITY:
Inclusion Criteria:

* > 55 years old
* admitted to one of the participating medical intensive care units (MICUs)
* intubated and on mechanical ventilation for acute respiratory failure
* expected to require mechanical ventilation for at least an additional 48 hours after enrollment.
* all critically ill patients age 55 and older with acute respiratory failure, on mechanical ventilation (invasive and noninvasive) or high flow oxygen therapy

Exclusion Criteria:

* coma due to structural brain diseases (e.g., stroke, intracranial hemorrhage, anoxic brain injury)
* expected death within 24 hours of study enrollment or lack of commitment to aggressive treatment by family/medical team
* inability to reach LAR to provide consent within 72 hours of ICU admission
* legal blindness or deafness because these patients cannot be assessed using the proposed study instruments
* airborne isolation precautions to minimize interventionists exposure and need for N95 respirators

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Establish the timing of subject recruitment | Days 1, 2, or 3
  Measured by the proportion of eligible patients enrolled on Days 1, 2, or 3 of mechanical ventilation initiation
Establish level of protocol adherence by participants | Days 1-5
  Measured by the number of days on protocol that subjects complete assigned intervention
Evaluate and refine the study protocol | Days 1-5
  Number of participants that complete the daily in-person pain, anxiety, and delirium assessments
Enrollment population | Days 1, 2, or 3
  Measured by the number and proportion of patients versus legally authorized representatives (LARs) who consent to study enrollment.
Establish level of protocol adherence by Interventionists | Days 1-5
  The ability of Reiki and sham Reiki interventionists to adhere to study protocol.
Facilitators/Barriers to successful Reiki Intervention implementation | Days 1-5
  Measure subject and LAR perception of the enrollment process, interventions, and symptom management effectiveness over the 5 day intervention period as assessed by the questionnaires completed .

SECONDARY OUTCOMES:
Pain assessed by numeric rating scale, (NRS) | Days 1-10
  Incidence, severity, and duration of pain as measured using a 0-10 visually enlarged horizontal pain numeric rating scale (NRS) in participants that can self report.
Pain assessed by Critical-Care Pain Observation Tool (CPOT) | Days 1-10
  Incidence, severity, and duration of pain as measured by the Critical-Care Pain Observation Tool (CPOT) for participants that are unable to self report. The CPOT has four behavioral categories: facial expression; body movements; muscle tension; and compliance with the ventilator for intubated subjects or vocalization for extubated subjects. Items in each section are scored 0 to 2, with a possible total score of 0 to 8.
Level of Arousal | Days 1 - 10
  As measured by Richmond Agitation and Sedation Scale (RASS) which is a 10-point scale, with four levels of anxiety or agitation ranging from +1 (restless) to +4 (combative), one level representing an alert and calm state (0), and five levels of sedation ranging from -5 (unarousable) to -1 (drowsy).
Delirium/ Coma free days | Days 1 - 10
  As measured by Confusion Assessment Method ICU (CAM-ICU) which includes four features of delirium: (1) acute onset or fluctuating course; (2) inattention; (3) disorganized thinking.
Anxiety level assessed with the Visual Analog Scale-Anxiety (VAS-A) | Days 1 - 10
  Anxiety will be measured with the 100-mm Visual Analog Scale-Anxiety. The VAS-A will be presented to participants with a vertical orientation; the bottom of the scale anchored by the statement "not anxious at all" and the top anchored by "most anxious ever." Subjects will indicate their current level of anxiety in response to the question "How anxious are you feeling today?"
Other symptoms | Days 1 - 10
  As measured by Patient Symptom Survey

CONTACTS AND LOCATIONS:
Overall Officials: Michele Balas, PhD, RN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No